CLINICAL TRIAL: NCT05957029
Title: Evaluation of Thermal Outcome and Safety of Nuera Tight RF System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LUM-VBU-NUERA-23-02
Record Dates: First submitted 2023-06-21; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-06

CONDITIONS: To Verify Tissue Heating and Temperature Stability and Safety Throughout RF Treatment Duration Applied on the Face

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Nuera Tight RF System (Experimental): Subjects will receive an RF treatment session on the periorbital area and cheeks with a frequency of 1 and 4 MHz. Each subject will be treated on one side of the face using a 10 mm capacitive electrode, and on the other side using a 20 mm capacitive electrode. The target temperature will be set at 42 C.
  Interventions: Device: NuEra Tight RF system

INTERVENTIONS:
Device: NuEra Tight RF system — monopolar radiofrequency device

SUMMARY:
The purpose of the study is to verify tissue heating, temperature stability and safety of the Nuera Tight RF device during and after treatment session applied on the face.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of either gender, 18 years of age or older
* Subject is able to read, understand and sign an informed consent form
* Subject is willing to comply with all study procedures

Exclusion Criteria:

* Subjects taking medicines that increase skin sensitivity to heat
* Subjects taking medicines that change skin metabolism
* Cancer or any pigmentary or vascular lesions in the planned treatment area
* Subjects with Herpes simplex in the area to be treated
* Pregnant women
* Subjects wearing pacemakers and/or any other type of implanted electronics
* Subjects with any inflammatory skin conditions
* Subjects with active cold sores, open lacerations, abrasions
* Chronic or acute skin infections
* Subjects with active local or systemic infections
* Subjects with any disease in which an increase of skin temperature is contraindicated
* Subjects wearing piercing in the area to be treated
* Subjects have nerve insensitivity to heat in the area to be treated
* Subjects have metal implants in the area to be treated, excluding dental implants
* Subjects allergic to glycerin, paraffin, parfum, parabens, nuts, vegetable oils, calendula, or chamomile
* Any condition where the study investigator determined that the subject is not adequate for this study
* Subjects participating in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
tissue heating | 12 minutes
  To verify tissue heating throughout the treatment duration applied on the face. The temperature will be set at 42 C, the operator will move the electrode in a continuous motion until the skin temperature reached the target temperature, then the treatment will continue for another 12 minutes. the skin temperature will be measured using an infrared thermometer to verify tissue heating
temperature stability | 12 minutes
  To verify temperature stability throughout the treatment duration applied on the face. the skin temperature will be measured using an infrared thermometer every 3 minutes to verify temperature stability

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lewis, MD, Principal Investigator — Lewis Dermatology & Associates; Shauna Diggs, MD, Principal Investigator — Cosmedic Dermatology
Locations (2):
- United States (2):
  - Cosmedic Dermatology, Detroit, Michigan
  - Lewis Dermatology & Associates, New York, New York

IPD SHARING:
Plan to Share IPD: No